CLINICAL TRIAL: NCT00128518
Title: IDEAL Study : Identification of the Determinants of the Efficacy of Arterial Blood Pressure Lowering Drugs
Brief Title: IDEAL Study: Identification of the Determinants of the Efficacy of Arterial Blood Pressure Lowering Drugs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2003.340
Record Dates: First submitted 2005-08-09; First posted 2005-08-10 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Hypertension
Keywords: Hypertension - Drugs - Blood pressure response - Responders - pharmacogenetics
MeSH Terms: conditions — Hypertension | interventions — Indapamide; Perindopril; P-2

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Group A : T1+P2 ● P1+P2 ● T2+P1 ● P1+P2 (Experimental): T1 = perindopril T2 = Indapamide P1 = Placebo of T1 P2 = Placebo of T2
  Interventions: Drug: Indapamide (T2); Drug: Perindopril (T1); Drug: Placebo of Perindopril (P1); Drug: Placebo of Indapamide (P2)
- Group B : P1+P2 ● T1+P2 ● P1+P2 ● T2+P1 (Experimental): T1 = perindopril T2 = Indapamide P1 = Placebo of T1 P2 = Placebo of T2
  Interventions: Drug: Indapamide (T2); Drug: Perindopril (T1); Drug: Placebo of Perindopril (P1); Drug: Placebo of Indapamide (P2)
- Group C : T2+P1 ● P1+P2 ● T1+P2 ● P1+P2 (Experimental): T1 = perindopril T2 = Indapamide P1 = Placebo of T1 P2 = Placebo of T2
  Interventions: Drug: Indapamide (T2); Drug: Perindopril (T1); Drug: Placebo of Perindopril (P1); Drug: Placebo of Indapamide (P2)
- Group D : P1+P2 ● T2+P1 ● P1+P2 ● T1+P2 (Experimental): T1 = perindopril T2 = Indapamide P1 = Placebo of T1 P2 = Placebo of T2
  Interventions: Drug: Indapamide (T2); Drug: Perindopril (T1); Drug: Placebo of Perindopril (P1); Drug: Placebo of Indapamide (P2)

INTERVENTIONS:
Drug: Indapamide (T2) — 1.5 mg/day during 4 weeks
Drug: Perindopril (T1) — 4 mg/day during 1 week then 8 mg/day during 3 weeks
Drug: Placebo of Perindopril (P1) — 1 pill/day during 1 week then 2 pills/day during 3 weeks
Drug: Placebo of Indapamide (P2) — 1 pill/day during 4 weeks

SUMMARY:
The principal scientific objective of the trial is to identify the factors that are associated with differential blood pressure responses between drugs. This may allow investigators to produce new hypotheses on the pathophysiology of hypertension and on the mechanisms of drug action.

These factors can be of different types:

* Environmental factors (sodium or alcohol intake);
* Morphological (height, weight, body mass index, body surface area);
* Initial blood pressure;
* Electrocardiogram (ECG) parameters of left ventricular hypertrophy;
* Biological parameters as the activity level of the renin angiotensin aldosterone system;
* Genetic polymorphisms.

ELIGIBILITY:
Inclusion Criteria:

* Participants have to be 25 to 60 years of age
* Both genders
* Systolic blood pressure of 140 mmHg or above; diastolic blood pressure of 90 mmHg or above.
* Cardiovascular risk must not be high, to allow for two periods of 4 weeks of placebo without ethical concern.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 139 (Actual)
Dates: Start 2004-10; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Blood pressure at the end of each 4 week treatment period | 16 weeks
  Change from baseline and after each 4 week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Francois GUEYFFIER, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Louis Pradel, Bron, France

REFERENCES:
- [Result] Gueyffier F, Subtil F, Bejan-Angoulvant T, Zerbib Y, Baguet JP, Boivin JM, Mercier A, Leftheriotis G, Gagnol JP, Fauvel JP, Giraud C, Bricca G, Maucort-Boulch D, Erpeldinger S; IDEAL Trial Group. Can we identify response markers to antihypertensive drugs? First results from the IDEAL Trial. J Hum Hypertens. 2015 Jan;29(1):22-7. doi: 10.1038/jhh.2014.29. Epub 2014 Apr 17. PMID 24739801